CLINICAL TRIAL: NCT06795009
Title: Phase I/IB Study of Zanzalintinib in Combination With Paclitaxel in Recurrent High Grade Uterine Cancer
Brief Title: Zanzalintinib in Combination With Paclitaxel in Recurrent High Grade Uterine Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202503049; P50CA265793 (NIH)
Record Dates: First submitted 2025-01-23; First posted 2025-01-27 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Uterine Cancer; Endometrial Cancer
Keywords: Recurrent endometrial cancer; AXL/GAS6; p53 mutation; High risk
MeSH Terms: conditions — Uterine Neoplasms; Endometrial Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 2 (Starting Dose): Zanzalintinib + Paclitaxel (Experimental): Patients will initiate paclitaxel on a 21-day cycle with the addition of zanzalintinib given on the same schedule. Dosing of zanzalintinib is dictated by the dose escalation schema. After 3 cycles, patients will be assessed for disease response. Patients who have progression will not continue on treatment. Patients who have a partial or complete response or stable disease will continue on treatment for another 3 cycles of paclitaxel + zanzalintinib at the assigned dose. Patients will be assessed for response again at the end of 6 cycles and may continue on treatment if they have partial response or stable disease. Up to 9 cycles of treatment with paclitaxel + zanzalintinib may be given. At the end of the 9 cycles, patients with a SD or PR can continue on maintenance zanzalintinib until progression. Patients with complete response after cycle 6 or 9 will continue single agent zanzalintinib as maintenance therapy until progression.
  Interventions: Drug: Zanzalintinib; Drug: Paclitaxel
- Dose Level 3: Zanzalintinib + Paclitaxel (Experimental): Patients will initiate paclitaxel on a 21-day cycle with the addition of zanzalintinib given on the same schedule. Dosing of zanzalintinib is dictated by the dose escalation schema. After 3 cycles, patients will be assessed for disease response. Patients who have progression will not continue on treatment. Patients who have a partial or complete response or stable disease will continue on treatment for another 3 cycles of paclitaxel + zanzalintinib at the assigned dose. Patients will be assessed for response again at the end of 6 cycles and may continue on treatment if they have partial response or stable disease. Up to 9 cycles of treatment with paclitaxel + zanzalintinib may be given. At the end of the 9 cycles, patients with a SD or PR can continue on maintenance zanzalintinib until progression. Patients with complete response after cycle 6 or 9 will continue single agent zanzalintinib as maintenance therapy until progression.
  Interventions: Drug: Zanzalintinib; Drug: Paclitaxel
- Dose Level 1 (Reduction): Zanzalintinib + Paclitaxel (Experimental): Patients will initiate paclitaxel on a 21-day cycle with the addition of zanzalintinib given on the same schedule. Dosing of zanzalintinib is dictated by the dose escalation schema. After 3 cycles, patients will be assessed for disease response. Patients who have progression will not continue on treatment. Patients who have a partial or complete response or stable disease will continue on treatment for another 3 cycles of paclitaxel + zanzalintinib at the assigned dose. Patients will be assessed for response again at the end of 6 cycles and may continue on treatment if they have partial response or stable disease. Up to 9 cycles of treatment with paclitaxel + zanzalintinib may be given. At the end of the 9 cycles, patients with a SD or PR can continue on maintenance zanzalintinib until progression. Patients with complete response after cycle 6 or 9 will continue single agent zanzalintinib as maintenance therapy until progression.
  Interventions: Drug: Zanzalintinib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Zanzalintinib — Taken by mouth.
  Other Names: XL092
Drug: Paclitaxel — 175 mg^m2 intravenous over 3 hours.
  Other Names: Taxol

SUMMARY:
The purpose of this study is to determine the recommended Phase 2 dose of zanzalintinib when given in combination with paclitaxel in patients with recurrent high-grade uterine cancer. Other objectives include overall safety and tolerability as well as rates of response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent, FIGO grade 3 endometrioid, serous, or mixed high grade uterine or endometrial cancer or uterine carcinosarcoma. Patients must have experienced either prior progression on a platinum-based therapy or intolerance to platinum. Patients with dMMR or MSI-H tumors or targetable HER2 alterations are required to have received prior therapy with appropriate targeted agents.
* 1-2 prior lines of anti-cancer therapy are allowed.
* Subjects who have received prior treatment with trastuzumab, pembrolizumab, or dostarlimab can enroll in the study. Use of these agents together or as maintenance therapy is considered 1 regimen.
* Recovery to baseline or ≤ Grade 1 severity (CTCAE v5) from adverse events (AEs), including immune-related adverse events (irAEs), related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy (eg, physiological replacement of corticosteroid). Low-grade or controlled toxicities such as alopecia, ≤ Grade 2 hypomagnesemia, ≤ Grade 2 neuropathy are permitted)
* Patients must have disease that cannot be managed by local therapy targeted at the tumor site (i.e. surgery, radiation therapy).
* Measurable disease by RECIST 1.1.
* At least 18 years of age.
* ECOG performance status ≤ 2.
* Adequate bone marrow and organ function within 14 days prior to first dose of study treatment, as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm without granulocyte colony-stimulating factor support within 2 weeks of screening laboratory sample collection.
  * Platelets ≥ 100 K/cumm ) without transfusion within 2 weeks of screening laboratory sample collection.
  * Hemoglobin ≥ 9.0 g/dL without transfusion within 2 weeks prior to screening laboratory sample collection.
  * Total bilirubin ≤ 1.5 x IULN (for subjects with Gilbert's disease ≤ 3 x ULN).
  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x ULN. For subjects with documented bone metastasis ALP ≤ 5 x ULN. Serum creatinine < 1.5 x ULN OR calculated or measured creatinine clearance ≥ 40 mL/min (using Cockcroft-Gault equation)
  * INR ≤ 1.5 x IULN
  * aPTT ≤ 1.2 x IULN
  * Urine protein-to-creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol) creatinine
* Female subjects of child-bearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria is met: permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating hormone [FSH] level > 40 mIU/mL to confirm menopause). Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff. Should a patient become pregnant or suspect pregnancy while participating in this study, the treating physician must be informed immediately.
* The effects of zanzalintinib on the developing human fetus are unknown. For this reason and because chemotherapeutic agents are known to be teratogenic, patients of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and through 186 days after last dose of zanzalintinib or paclitaxel for women of child-bearing potential (WOCBP). An additional contraceptive method, such as a barrier method (eg, condom), is required. In addition, women must agree not to donate eggs (ova, oocyte) for the purpose of reproduction during these same periods.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Any prior treatment with zanzalintinib
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease.
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment, or any prior treatment with any tyrosine kinase inhibitor (TKI) or any prior treatment with bevacizumab.
* Receipt of any other (non-study) cytotoxic chemotherapy, radiation, targeted treatment, or immunotherapy (including investigational) within 4 weeks prior of start of study treatment.
* Receipt of any other investigational agents or has received an investigational agent within 4 weeks of start of study treatment.
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Note: Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of enrollment. Note: Base of skull lesions without definitive evidence of dural or brain parenchymal involvement are allowed.
* Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin inhibitors ) and platelet inhibitors (eg, clopidogrel).

  * Allowed anticoagulants are the following:

    * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
    * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen. Note: Subjects must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to first dose of study treatment, whichever is longer.
* Any complementary medications (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before first dose of study treatment.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Unstable or deteriorating cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class 3 or 4, class 2 or higher, unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (eg, ventricular flutter, ventricular fibrillation, Torsades de pointes).
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant arterial thrombotic and/or ischemic event within 6 months before first dose of study treatment.
    * Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous events within 3 months before first dose of study treatment. Note: Subjects with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen. Note: Subjects who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the Principal Investigator.
    * Prior history of myocarditis.
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * Tumors invading the GI-tract from external viscera
    * Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis
    * Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months before first dose unless cause of obstruction is definitively managed and subject is asymptomatic
    * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
    * Known gastric or esophageal varices
    * Ascites, pleural effusion, or pericardial fluid requiring drainage in last 4 weeks
    * If tolerating PO, small bowel obstruction may be considered with Investigator and Sponsor approval
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
* Symptomatic cavitating pulmonary lesion(s) or endobronchial disease (asymptomatic or radiated lesions allowed).
* Lesions invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta.
* Other clinically significant disorders that would preclude safe study participation.

  * Active infection requiring systemic treatment. Note: Prophylactic antimicrobial treatments (antibiotics, antimycotic, antiviral) are allowed.
  * Known infection with acute or chronic hepatitis B or C, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness except for subjects meeting all of the following criteria: (1) on stable anti-retroviral therapy; (2) CD4+ T cell count ≥ 200/µL; and (3) an undetectable viral load. Note: HIV testing will be performed at screening if and as required by local regulation. Note: To be eligible, participants taking CYP inhibitors (eg, zidovudine, ritonavir, cobicistat, didanosine) or CYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies (ART) must have been received for at least 4 weeks prior to the first dose. Note: CD4+ T cell counts, and viral load are monitored per standard of care by the local health care provider.
  * Serious non-healing wound/ulcer/bone fracture. Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.
  * Malabsorption syndrome.
  * Pharmacologically uncompensated, symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
  * Requirement for hemodialysis or peritoneal dialysis.
  * History of solid organ or allogeneic stem cell transplant.
* Major surgery within 8 weeks prior to first dose of study treatment. Prior laparoscopic surgeries (ie nephrectomy) within 4 weeks prior to first dose of study treatment. Minor surgery (eg, simple excision, tooth extraction) within 5 days before first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to first dose of study treatment. Note: Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms within 14 days per electrocardiogram (ECG) before first dose of study treatment. Note: Triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.
* History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
* Pregnant or lactating females.
* Inability to swallow tablets
* Previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Another malignancy that requires active therapy and in the opinion of the Investigator would interfere with monitoring of radiologic assessments of response to Investigational Product, within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy.
* Other conditions, which in the opinion of the Investigator, would compromise the safety of the patient or the patient's ability to complete the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2035-04-30 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 dose (RP2D) | Through completion of first cycle (each cycle is 21 days) of all enrolled patients (estimated to be 48 months and 3 weeks)

SECONDARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events | From start of treatment through 30 days after last dose of zanzalinitinib (estimated to be 7 months)
Overall response rate (ORR) | After 3 cycles of treatment (each cycle is 21 days - estimated to be 63 days)
  ORR is defined as the proportion of subjects who have a partial or complete response per RECIST criteria after 3 cycles of treatment with zanzalintinib plus paclitaxel.
Progression-free survival (PFS) | From start of treatment through completion of follow-up (estimated to be 5.5 years)
  PFS is defined as the time from start of treatment to the first radiologically documented disease progression, or death, whichever comes first. The alive patients without radiologically documented disease progression are censored at the last follow-up.
Overall survival (OS) | From start of treatment through completion of follow-up (estimated to be 5.5 years)
  OS is defined as the time from start of treatment to death. The alive patients are censored at the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: David G Mutch, M.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - University of California, San Francisco, San Francisco, California
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Oklahoma, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu